CLINICAL TRIAL: NCT06972134
Title: Synergistic Effects of Sesame Oil, Extra Virgin Olive Oil, Psyllium Extract, and Dandelion Extract on Cholesterol Gallstone Dissolution: An In Vitro Comparative Study Against Rowachol®
Brief Title: Synergistic Effects of Natural Oils and Herbal Extracts on Cholesterol Gallstone Dissolution: In Vitro Comparison With Rowachol®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Duhok (Other)
Responsible Party: Principal Investigator, Mohamad Radwan Sirri, Clinical Professor, University of Duhok
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIU-618-11GR-1358; AIU-618-11GR (Registry Identifier: AIU-618-11GR)
Record Dates: First submitted 2025-04-28; First posted 2025-05-14 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Cholesterol Gallstone Dissolution
Keywords: Gallstone dissolution; Cholesterol gallstones; Natural oils; Herbal extracts; Oleic Acid; Taraxacin; Rowachol®; In vitro study
MeSH Terms: interventions — Sesame Oil; Olive Oil; Psyllium; Rowachol; Terpenes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Group 1 (G1) (Experimental): Sesame oil (SO) at 100 mg/mL in dissolving fluid.
  Interventions: Dietary Supplement: Sesame Oil (SO) at 100 mg/mL in dissolving fluid.
- Group 2 (G2) (Experimental): Extra Virgin Olive Oil (EVOO) at 100 mg/mL in dissolving fluid.
  Interventions: Dietary Supplement: Extra Virgin Olive Oil (EVOO) at 100 mg/mL in dissolving fluid.
- Group 3 (G3) (Experimental): 50% Sesame Oil + 50% Extra virgin Olive Oil.
  Interventions: Dietary Supplement: 50% Sesame Oil (SO) + 50% Extra Virgin Olive Oil (EVOO).
- Group 4 (G4) (Experimental): 50% Psyllium + 50% Oils (a mixture of 50% Sesame Oil + 50% Extra virgin Olive Oil).
  Interventions: Dietary Supplement: 50% Psyllium Extract (PE) + 50% Oil Blend (50% SO + 50% EVOO).
- Group 5 (G5) (Experimental): : 50% Dandelion + 50% Oils (a mixture of 50% Sesame Oil + 50% Extra virgin Olive Oil).
  Interventions: Dietary Supplement: Plantago ovata extract (AIU-BC-618-4) + AIU-BC-618-3
- Group 6 (G6) (Experimental): 50% Herbal extract (50% Dandelion + 50% Psyllium) + 50% Oils (a mixture of 50% 50% Sesame Oil + 50% Extra virgin Olive Oil).
  Interventions: Dietary Supplement: 50% Herbal Extract (25% PE + 25% DE) + 50% Oil Blend (25% SO + 25% EVOO).
- Group 7 (G7) - Control (Active Comparator): Rowachol® (terpene extract) at 100 mg/mL in dissolving fluid.
  Interventions: Drug: Drug: Rowachol® (terpene extract) at 100 mg/mL in dissolving fluid.

INTERVENTIONS:
Dietary Supplement: Sesame Oil (SO) at 100 mg/mL in dissolving fluid. — Pure Sesamum indicum oil (cold-pressed, unrefined) dissolved in BioIVT bile juice at 100 mg/mL. Prepared by homogenization (30 min, 37°C). Used as monotherapy.
  Other Names: Sesamum indicum oil (AIU-BC-618-1)
  Arms: Group 1 (G1)
Dietary Supplement: Extra Virgin Olive Oil (EVOO) at 100 mg/mL in dissolving fluid. — Pure Olea europaea oil (first cold-pressed, acidity ≤0.8%) dissolved in BioIVT bile juice at 100 mg/mL. Prepared by vortex mixing (15 min, 25°C). Used as monotherapy.
  Other Names: Olea europaea oil (AIU-BC-618-2)
  Arms: Group 2 (G2)
Dietary Supplement: 50% Sesame Oil (SO) + 50% Extra Virgin Olive Oil (EVOO). — A 1:1 (v/v) blend of Sesamum indicum oil (AIU-BC-618-1) and Olea europaea oil (AIU-BC-618-2). Final concentration: 100 mg/mL in BioIVT bile juice. Prepared by mechanical stirring (1 hr, 40°C).
  Other Names: AIU-BC-618-3 (Synergistic Oil Blend)
  Arms: Group 3 (G3)
Dietary Supplement: 50% Psyllium Extract (PE) + 50% Oil Blend (50% SO + 50% EVOO). — 50% Plantago ovata mucilage extract (aqueous extraction, 65°C) + 50% AIU-BC-618-3 (SO+EVOO blend). Final concentration: 100 mg/mL in BioIVT bile juice. Prepared by sonication (20 min).
  Other Names: Plantago ovata extract (AIU-BC-618-4) + AIU-BC-618-3
  Arms: Group 4 (G4)
Dietary Supplement: Plantago ovata extract (AIU-BC-618-4) + AIU-BC-618-3 — 50% Taraxacum officinale root extract (ethanol-water extraction, 70°C) + 50% AIU-BC-618-3 (SO+EVOO blend). Final concentration: 100 mg/mL in BioIVT bile juice. Prepared by magnetic stirring (30 min, 50°C).
  Other Names: Taraxacum officinale extract (AIU-BC-618-5) + AIU-BC-618-3
  Arms: Group 5 (G5)
Dietary Supplement: 50% Herbal Extract (25% PE + 25% DE) + 50% Oil Blend (25% SO + 25% EVOO). — 25% Plantago ovata extract (AIU-BC-618-4) + 25% Taraxacum officinale extract (AIU-BC-618-5) + 25% SO (AIU-BC-618-1) + 25% EVOO (AIU-BC-618-2). Final concentration: 100 mg/mL in BioIVT bile juice. Prepared by homogenization (45 min, 37°C).
  Other Names: AIU-BC-618-6 (Full Synergy Formulation)
  Arms: Group 6 (G6)
Drug: Drug: Rowachol® (terpene extract) at 100 mg/mL in dissolving fluid. — 25% Plantago ovata extract (AIU-BC-618-4) + 25% Taraxacum officinale extract (AIU-BC-618-5) + 25% SO (AIU-BC-618-1) + 25% EVOO (AIU-BC-618-2). Final concentration: 100 mg/mL in BioIVT bile juice. Prepared by homogenization (45 min, 37°C).
  Other Names: Rowachol® (A. Nattermann & Cie. GmbH, Germany; FDA NDC 12345-678-90; Batch No. ROW-2024-SYR)
  Arms: Group 7 (G7) - Control

SUMMARY:
Objective:

This study aims to evaluate the effectiveness of a natural mixture (sesame oil, extra virgin olive oil, psyllium extract, and dandelion extract) in dissolving cholesterol gallstones compared to the standard medication, Rowachol®.

Methods:

In laboratory experiments, 70 cholesterol gallstones obtained from 55 patients were divided into seven groups. Each group was treated with different combinations of the natural ingredients or Rowachol®. The stones were monitored for 144 hours to measure dissolution rate and cholesterol release.

ELIGIBILITY:
Inclusion Criteria:

----------------------------------- Diagnosis of cholesterol gallstones requiring surgical removal. Gallstones with ≥70% cholesterol composition (confirmed via FTIR). Gallstone size: 10-13 mm (measured via digital caliper). Gallstone weight: 120-150 mg (measured via electronic balance). Age range: 40-50 years. BMI: 20-30 kg/m².

------------------------------------------------------------------------------------------------------------------------------

Exclusion Criteria:

----------------------------------- Hepatitis B/C infection. Chronic or acute illnesses (e.g., liver cirrhosis, hemolytic anemia). Pregnancy or lactation. History of malignancy. Participation in other clinical trials within the past 3 months.

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Gallstone Dissolution Rate | 48-hours, 96-hours, 144 hours
  Percentage reduction in gallstone weight after treatment.
  Calculated using the formula:
  DR%= (W initial-W final)/ W initial×100 Measurement Tool: Ohaus Adventurer Pro AV-2102 balance Unit of Measure: %
Cholesterol Release | 48-hours, 96-hours, 144 hours
  Total cholesterol released from gallstones into the dissolving medium. Measurement Tool: Cholestech LX-20 autoanalyzer Unit of Measure: mg

SECONDARY OUTCOMES:
Bioactive Compound Concentration | Baseline (T0)
  Quantification of key compounds (oleic acid, taraxacin, arabinoxylan, linoleic acid) in treatment solutions.
  Measurement Tool: GC-MS (fatty acids), HPLC (plant extracts) Unit of Measure: mg/mL
Synergistic Interaction Efficacy | 144 hours (T3)
  Comparative analysis of dissolution rates and cholesterol release between combined and individual treatments.
  Measurement Tool: Ohaus Balance + Cholestech LX-20 Unit of Measure: %, mg
Correlation: Compounds vs. Outcomes | 144 hours (T3)
  Pearson correlation coefficients between bioactive compound concentrations and dissolution metrics.
  Measurement Tool: Statistical analysis (SPSS v26) Unit of Measure: r-value (unitless)
Predictive Factors of Dissolution | 144 hours (T3)
  Multiple regression analysis identifying key predictors (e.g., oleic acid, taraxacin) of efficacy.
  Measurement Tool: Statistical analysis (SPSS v26) Unit of Measure: β-coefficient

CONTACTS AND LOCATIONS:
Locations (1):
- Arab International University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fan M, Zhang X, Song H, Zhang Y. Dandelion (Taraxacum Genus): A Review of Chemical Constituents and Pharmacological Effects. Molecules. 2023 Jun 27;28(13):5022. doi: 10.3390/molecules28135022. PMID 37446683
- [Background] Kumar, Pandey J, Kumar P, et al.; Psyllium Mucilage and Its Use in Pharmaceutical Field: An Overview. Current Synthetic and Systems Biology 2017;05. doi: 10.4172/2332-0737.1000134.
- [Background] Zommara MA, Swelam S, Raya-Alvarez E, Imaizumi K, Elmahdy A, Alkhudhayri DA, Aljehani AA, Agil A, Elmahallawy EK. Nutritional and potential health benefits of chufa oil, olive oil, and anhydrous milk fat against gallstone disease in a C57BL/6N mouse model. Front Nutr. 2024 Sep 26;11:1445484. doi: 10.3389/fnut.2024.1445484. eCollection 2024. PMID 39391681
- [Background] Vahedi H, Atefi M, Entezari MH, Hassanzadeh A. The effect of sesame oil consumption compared to sunflower oil on lipid profile, blood pressure, and anthropometric indices in women with non-alcoholic fatty liver disease: a randomized double-blind controlled trial. Trials. 2022 Jul 8;23(1):551. doi: 10.1186/s13063-022-06451-1. PMID 35804451
- [Background] Stokes CS, Gluud LL, Casper M, Lammert F. Ursodeoxycholic acid and diets higher in fat prevent gallbladder stones during weight loss: a meta-analysis of randomized controlled trials. Clin Gastroenterol Hepatol. 2014 Jul;12(7):1090-1100.e2; quiz e61. doi: 10.1016/j.cgh.2013.11.031. Epub 2013 Dec 7. PMID 24321208